CLINICAL TRIAL: NCT05891821
Title: Assessment of the Safety and Efficacy of Balstilimab for the Treatment of Relapsed/Refractory Lymphomas (IMMONC0001)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immune Oncology Research Institute (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMONC0001
Record Dates: First submitted 2023-05-11; First posted 2023-06-07 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Balstilimab (Experimental): 300 mg IV every 3 weeks for a maximum of 24 months
  Interventions: Drug: Balstilimab

INTERVENTIONS:
Drug: Balstilimab — An anti-programmed death (ligand) 1 [PD-(L)1] monoclonal antibody
  Other Names: AGEN2034

SUMMARY:
The goal of this study is to see if the drug balstilimab is safe and effective in participants with relapsed/refractory lymphomas.

Participants will receive balstilimab every 3 weeks and their outcomes will be assessed periodically.

DETAILED DESCRIPTION:
This is a single-arm, open-label phase 2 study to evaluate the safety and efficacy of single agent balstilimab in participants with relapsed/refractory lymphoma. The study will enroll participants with relapsed/refractory classical Hodgkin lymphoma or primary mediastinal B-cell lymphoma. The participants will receive balstilimab (BAL) 300 mg IV every 3 weeks. BAL infusions will be administered within 30 minutes (± 5 min) using an infusion pump.

The total estimated maximum time of study participation for each patient is approximately 49 months across 3 periods:

* Screening Period: approximately 28 days
* Treatment Period: up to 24 months, or until any criterion for stopping the study drug or withdrawal from the study occurs
* Follow-up Period: up to 24 months from last dose of study treatment for every patient who is alive

Study Duration

* Recruitment: 2 years
* Treatment: 2 years
* Follow-up: 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate by giving written informed consent
2. ≥ 18 years of age
3. Have a histologically confirmed diagnosis of a relapsed/refractory classical Hodgkin lymphoma (cHL) or primary mediastinal B-cell lymphoma (PMBCL) for which no standard therapy is available or standard therapy has failed or the patient does not have access to it.
4. Has a life expectancy of at least 3 months and an ECOG performance status of ≤1 as determined by study Investigator
5. Patients must have sufficient and adequate formalin-fixed tumor tissue sample available that is not older than 3 years; otherwise, a fresh biopsy is required. Archival tissue or fresh biopsy must be from a site not previously irradiated
6. Has adequate organ function defined as the following laboratory values within 7 days of C1D1:

   1. Neutrophils ≥ 1500/μL (Must be stable and off any growth factor within 4 weeks of first study treatment administration)
   2. Platelets ≥ 75 × 103/μL (transfusion to achieve this level is not permitted within 2 weeks of first study treatment administration)
   3. Hemoglobin ≥ 8.0 g/dL (transfusion to achieve this level is not permitted within 2 weeks of first study treatment administration)
   4. Creatinine clearance ≥ 30 mL/min as measured or calculated per local institutional standards
   5. AST/ALT ≤ 3 × upper limit of normal (ULN)
   6. Total bilirubin ≤ 1.5 × ULN (except patients with Gilbert syndrome who must have a total bilirubin level of ≤ 3.0 × ULN)
7. Women of childbearing potential (WOCP) must have a negative serum pregnancy test at Screening (within 7 days before first dose of study drug). Non-childbearing potential is defined as (by other than medical reasons):

   1. ≥ 50 years of age and has not menstruated for greater than 1 year
   2. Whose status is post hysterectomy, bilateral oophorectomy, or tubal ligation
   3. WOCP must be willing to use highly effective methods of contraception (defined in the informed consent form [ICF]) throughout the study, starting with the Screening Visit through 90 days after the last dose of study drug Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
8. Male patients with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the study starting with the screening visit through 90 days after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.
9. Is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

1. Has an inadequate period of time prior to first dose of study treatment that is defined as:

   1. Received systemic cytotoxic chemotherapy within 3 weeks before initiation of study treatment
   2. Received biological therapy or investigational therapy within 4 weeks or 5 circulating halve-lives, whichever is shorter
   3. Received small molecule/tyrosine kinase inhibitors within 2 weeks or 5 circulating half-lives, whichever is shorter
   4. Received radiation therapy within 3 weeks before initiation of study treatment, except for palliative radiation therapy, which can be received 2 weeks prior to initiation of study treatment
   5. Had major surgery within 4 weeks before initiation of study treatment
2. Has gone through disease progression after receiving prior therapy with:

   a. Any antibody/drug targeting T-cell co-regulatory proteins (immune checkpoints) such as anti-PD-1 and anti-PD-L1 antibodies
3. Has persisting AEs related to prior immunotherapy of NCI-CTCAE v5.0 Grade ≥ 2 severity.
4. Is expected to require any other form of systemic or localized antineoplastic therapy while on study (including maintenance therapy with another agent, radiation therapy, and/or surgical resection)
5. Has known allergy or hypersensitivity to any component of balstilimab, any history of anaphylaxis, or uncontrolled asthma
6. Has active or history of autoimmune disease that requires systemic treatment within 2 years of the start of study drug (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs) Note: Patients with autoimmune conditions requiring hormone replacement therapy or topical treatments are eligible.
7. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses (≤ 10 mg daily prednisone equivalent) are permitted in the absence of active autoimmune disease.
8. Has had an allogeneic tissue/solid organ transplant
9. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ III), or serious uncontrolled cardiac arrhythmia requiring medication.

   a. QTcF (QTc interval corrected using Fridericia's formula) of > 480 ms.
10. Any evidence of current interstitial lung disease (ILD) or pneumonitis, or prior history of ILD or non-infectious pneumonitis requiring glucocorticoids.
11. Has known untreated hepatitis B/hepatitis C virus (HBV/HCV) or tuberculosis. Active HBV is defined as a known positive hepatitis B surface antigen result. Active HCV is defined by a known positive hepatitis C antibody result and known quantitative HCV RNA results greater than the lower limits of detection of the assay
12. Uncontrolled infection with human immunodeficiency virus (HIV). Patients on stable highly active antiretroviral therapy with undetectable viral load and normal CD4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required.
13. Has other systemic conditions or organ abnormalities that in the opinion of the Investigator may interfere with the conduct and/or interpretation of the current study
14. Has known psychiatric or substance use disorders that would interfere with cooperation or compromise participation with the requirements of the study
15. Is legally incapacitated or has limited legal capacity
16. Is pregnant or breastfeeding
17. Has received a live/attenuated vaccine within 14 days of first dose of study treatment and other vaccines within 48 hours of first dose of study treatment
18. Has other co-morbidities that would alter risk-benefit of providing balstilimab (determined by treating physician's assessment)
19. Is receiving other therapy that would alter risk-benefit of providing balstilimab (determined by treating physician's assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | First dose to up to 27 months
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) assessed per the Lugano criteria

SECONDARY OUTCOMES:
Duration of Response (DOR) | First dose to up to 27 months
  DOR is defined as time from first observation of response to first observation of documented disease progression per the Lugano criteria or death within 12 weeks of last tumor assessment
Disease Control Rate (DCR) | First dose to up to 27 months
  DCR is defined as the percentage of patients who have achieved complete response, partial response or stable disease per the Lugano criteria
Duration of Stable Disease (SD) | First dose to up to 27 months
  Duration of SD is measured from the start of treatment until the criteria for progression are met, per the Lugano criteria
Time to Response | First dose to up to 27 months
  Time to Response is defined as the time from the first dose date to first observation of confirmed response per the Lugano criteria
Progression-Free Survival (PFS) Time | First dose to up to 27 months
  PFS time is defined as time from first treatment administration to first observation of documented disease progression (or death within 12 weeks after last tumor assessment), per the Lugano criteria
Overall Survival (OS) Time | First dose to up to 48 months
  OS Time is defined as time from start of treatment to death
Baseline expression of PD-L1 association with ORR | First dose to up to 48 months
  Tumor PD-L1 status will be determined and correlation with ORR will be investigated
Baseline expression of PD-L1 association with DOR | First dose to up to 48 months
  Tumor PD-L1 status will be determined and correlation with DOR will be investigated
Baseline expression of PD-L1 association with PFS | First dose to up to 48 months
  Tumor PD-L1 status will be determined and correlation with PFS time will be investigated
Baseline expression of PD-L1 association with OS | First dose to up to 48 months
  Tumor PD-L1 status will be determined and correlation with OS time will be investigated
Frequency, severity, and duration of treatment emergent adverse events (TEAEs) and laboratory abnormalities | First dose to up to 27 months
  TEAEs are reported using the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Gevorg Tamamyan, MD, PhD, DSc, Study Director — Immune Oncology Research Institute; Samvel Bardakhchyan, MD, PhD, Study Chair — Immune Oncology Research Institute; Astghik Voskanyan, MD, Principal Investigator — Hematology Center named after Prof. R. Yeolyan
Locations (1):
- Hematology Center named after prof. R. Yeolyan, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No